CLINICAL TRIAL: NCT01523847
Title: A Phase II Multi-centre Study of MBVD in Elderly and/or Cardiopathic Patients Affected by Hodgkin's Lymphoma (HL)
Brief Title: A Multi-centre Study of MBVD in Elderly and/or Cardiopathic Patients Affected by Hodgkin's Lymphoma (HL)
Acronym: HD0803
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Collaborators: Centro di Riferimento per l'Epidemiologia e la Prev. Oncologica Piemonte (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIL - HD0803; EudraCT Number 2009-013839-37
Record Dates: First submitted 2011-06-22; First posted 2012-02-01 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Hodgkin Lymphoma
Keywords: Hodgkin Lymphoma; Cardiopathic; elderly; Myocet
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MBVD (Myocet+BVD) (Experimental): 2 MBVD courses, after early restaging with PET scan (PET-2)
  The subsequent treatment will be planned as follows:
  * -Stage I and IIA patients will go on with 1 more course of MBVD (total of 3 courses) followed by involved field radiotherapy (30 Gy-36 Gy).
  * -Advanced stage (IIB-IV) patients will go on with 4 more courses of MBVD (total of 6 courses). Radiotherapy limited to bulky or non complete responder areas (30 Gy) is optional.
  Interventions: Drug: MBVD (Myocet+BVD)

INTERVENTIONS:
Drug: MBVD (Myocet+BVD) — MBVD will be scheduled as follows:
  Myocet 25 mg/mq i.v. day 1 and 15 Bleomycin 10 mg/mq i.v. day 1 and 15 Vinblastine 6 mg/mq i.v. day 1 and 15 Dacarbazine 375 mg/mq i.v. day 1 and 15
  Other Names: MBVD

SUMMARY:
The study has the purpose to evaluate in elderly and/or cardiopathic HL patients, the cardiologic toxicity of the MBVD regimen, where liposomal doxorubicin (Myocet®) is substituted for doxorubicin in the conventional ABVD regimen.

DETAILED DESCRIPTION:
STUDY POPULATION Patients affected by Hodgkin's lymphoma, any stage, older than 69 years. Patients affected by Hodgkin's Lymphoma with concomitant cardiopaty, older than 18 years.

AIMS OF THE STUDY

* To evaluate in elderly and/or cardiopathic HL patients, the cardiologic toxicity of the MBVD regimen, where liposomal doxorubicin (Myocet®) is substituted for doxorubicin in the conventional ABVD regimen
* To compare in a pair-match retrospective analysis the results obtained with MBVD with those obtained in patients comparable for clinical variables and treated with ABVD or with the reduced intensity VEPEMB schedule.

STUDY DESIGN Multi-centre phase II study SAMPLE SIZE 50 patients

STUDY PROCEDURES

* Histologic diagnosis of Hodgkin Lymphoma.
* Early Staging evaluation including:

  * Blood tests
  * CT, PET and bone marrow biopsy.
  * Heart and lung function evaluation.
  * Geriatric assessment.
  * Quality of life evaluation.
* 2 MBVD courses
* Early restaging with PET scan (PET-2)
* The subsequent treatment will be planned as follows:

  * Stage I and IIA patients will go on with 1 more course of MBVD (total of 3 courses) followed by involved field radiotherapy (30 Gy-36Gy).
  * Advanced stage (IIB-IV) patients will go on with 4 more courses of MBVD (total of 6 courses). Radiotherapy limited to bulky or non complete responder areas (30-36 Gy) is optional.
* Final restaging including:

  * Blood tests
  * CT, PET
  * bone marrow biopsy if positive at baseline.
  * Heart and lung function evaluation.
  * Geriatric assessment.
  * Quality of life evaluation

Follow up procedures will include:

1. a clinical and laboratory evaluation (with troponin, proBNP / BNP, cardiology visit, ECG and echocardiogram) every 6 months in the first 2 years, then annually.
2. CT scans will be planned annually.
3. Compilation of geriatric evaluation scales every 6 months in the first 2 years, then annually.

MBVD will be scheduled as follows (4 weeks):

Myocet 25 mg/mq i.v. day 1 and 15 Bleomycin 10 mg/mq i.v. day 1 and 15 Vinblastine 6 mg/mq i.v. day 1 and 15 Dacarbazine 375 mg/mq i.v. day 1 and 15 Supportive treatment with G-CSF and/or Erythropoietin will be planned according to international guide-lines.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Hodgkin's lymphoma, except for nodular lymphocyte predominance subgroup.
* Previously untreated
* Age ≥ 70.
* Age> 18 in presence of cardiopathy according to inclusion criteria…
* Patients with HCV and HBV infection can be included. For patients HBV+ occult carriers (AntiHBc+, HbsAg-, AntiHBs+/-) Lamivudine prophylaxis is mandatory.
* Life expectancy >3 months
* Informed consent.
* Staging with PET-CT.
* Preliminary geriatric assessment (ADL, IADL, co-morbidity and frailness scores).

Exclusion Criteria:

* Lymphocyte predominance subgroup
* Age < 70 (no cardiopathy)
* Age < 18 (with cardiopathy).
* HIV infection.
* Previous treatments for Hodgkin's lymphoma.
* Other concomitant or previous malignancies, with the exception of basal cell skin tumors, adequately treated carcinoma in situ of the cervix and any cancer that has been in complete remission for > 5 years.
* Renal failure (creatinine higher than twice the normal level) or liver disease (AST/ALT or bilirubin level higher than 2.5 times the normal level)
* Other clinical situations that contraindicate, to the judgment of investigators, the administration of a mild-dose chemotherapy. Isolated comorbidities will be scored and recorded, but they are not, if isolated, a sufficient reason for exclusion.
* Frail patients, defined according to comorbidity scale: patients with 1 grade 4 comorbidity, or >3 grade 3 comorbidities, are excluded. (see appendix.6)
* Unresponsive sepsis
* Dementia
* Impossibility to subscribe the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Complete Response (CR) at the end of the chemotherapy program | 24 weeks
  CR is defined according to the Cheson 2007 response criteria.
Cardiac Toxicity during the chemotherapy program measured by CTCAE v.3 | 24 weeks
  Evaluation of Cardiac Toxicity during the chemotherapy program measured by CTCAE v.3

SECONDARY OUTCOMES:
Cardiac toxicity of MBVD after two courses of MBVD measured by CTCAE v.3 | 8 weeks
  Evaluation of cardiac toxicity of MBVD in elderly and/or cardiopathic patients with Hodgkin's lymphoma after two courses of MBVD.
Progression Free Survival (PFS) | 24 months
  PFS will be measured from the day of enrolment to the date of disease progression, relapse or death due to any cause
Relapse Free Survival (RFS) of patients entering complete remission | 24 months
  RFS is defined only for patients who achieve CR, and is measured from the date of attaining the disease-free state until the date of relapse or death from any cause
Overall Survival (OS) | 24 months
  OS will be measured from the day of enrolment to the date of relapse or death due to any cause
Change from the theoretical total amount of drug delivered in a one-week period (dose-intensity) | 24 weeks
  Proportion of dose-intensity delivered to patients
Change in cardiac markers during and at the end of chemotherapy | 24 weeks
  Evaluate Change in cardiac markers during and at the end of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Levis, PhD, Study Director — Azienda Ospedaliera SS Antonio, Biagio e Cesare Arrigo
Locations (26):
- Italy (26):
  - Azienda Ospedaliera SS. Antonio e Biagio e C. Arrigo, Alessandria, Alessandria
  - Ospedale "A. Perrino", Brindisi, Brindisi
  - Ematologia Ospedale Vito Fazzi, Lecce, Lecce
  - Ospedale Cardinale Giovanni Panico, Tricase, Lecce
  - A.S.U.R. Zona Territoriale n°8 - Ospedale di Civitanova Marche U.O. Medicina Interna ed Ematologia, Civitanova Marche, Macerata
  - Azienda Ospedaliera V.Cervello, Palermo, Palermo
  - Ospedale Guglielmo da Saliceto, Piacenza, Piacenza
  - Azienda Ospedaliera "Bianchi Melacrino Morelli", Reggio Calabria, Reggio Calabria
  - Ematologia Azienda Ospedaliera Arcispedale "S. Maria Nuova", Reggio Emilia, Reggio Emilia
  - Divisione di Oncologia Ospedale civile degli Infermi, Rimini, Rimini
  - U.O.C. Ematologia IRCCS Istituti Fisioterapici Ospitalieri, Roma, Roma
  - SC Medicina trasfusionale ed Ematologia Ospedale civile di Ivrea, Ivrea, Torino
  - Struttura Complessa di Ematologia PO TREVISO, Treviso, Treviso
  - Centro di riferimento Oncologico, Aviano
  - IRCC Istituto Tumori, Bari
  - Policlinico S. Orsola Malpighi, Bologna
  - Spedali Civili, Brescia
  - Ospedale Businco, Cagliari
  - Area Vasta Romagna e IRST, Meldola (FC)
  - Ospedale Maggiore della Carità, Novara
  - Fondazione Policlinico San Matteo, Pavia
  - Osp. S. Maria delle Croci, Ravenna
  - Ospedale S. Eugenio, Roma
  - Università "La Sapienza", Roma
  - Ospedale Santa Maria, Terni
  - Azienda Ospedaliero - Universitaria di Udine, Udine